CLINICAL TRIAL: NCT05141994
Title: Phase II Clinical Study on the Efficacy and Safety of BAT5906 Injection in the Vitreous Age-related Macular Degeneration Patients With Two Repeated Intravitreal Dose
Brief Title: Clinical Study on the Efficacy and Safety of BAT5906 Injection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAT5906-002-CR
Record Dates: First submitted 2020-06-22; First posted 2021-12-02 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Wet Age-related Macular Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2.5mg of BAT5906 (Experimental): Specification: 10mg/0.2ml/piece; route: intravitreal injection; dose: 2.5mg/eye/time, 50μl; medication duration: about once every 4 weeks, taking 3 times after continuous use, effective observation to Week 48.
  Interventions: Drug: 2.5mg of BAT5906
- 4.0mg of BAT5906 (Experimental): 16mg/0.2ml/piece; route of administration: intravitreal injection; dose: 4.0mg/eye/time, 50μl; duration of administration: once every 4 weeks, 3 times after continuous administration , The effectiveness was observed to the 48th week.
  Interventions: Drug: 4mg of BAT5906

INTERVENTIONS:
Drug: 2.5mg of BAT5906 — Specification: 2.5mg of BAT5906
  Arms: 2.5mg of BAT5906
Drug: 4mg of BAT5906 — Specification: 4mg of BAT5906
  Arms: 4.0mg of BAT5906

SUMMARY:
This study is a multi-center, open, and phase II clinical study to evaluate the efficacy and safety of BAT5906 injection in patients with wet age-related macular degeneration. The results of the BAT5906 Phase I study show that it is safe from 0.3-4.0 mg, and that higher doses (2.5 mg and 4 mg) may be substituted for the duration of maintenance efficacy; drugs with the same target (such as brolucizumab and Abecip) have also been found in clinical studies High doses can extend the interval and reduce the frequency of administration. Therefore, in this study, two doses with better safety and efficacy were selected, once every 4 weeks, followed by 3 consecutive injections for treatment as needed, and preliminary exploration of the best clinical effective dose and replacement frequency

ELIGIBILITY:
Inclusion Criteria:

* Only the following criteria are met:

  1. The patient or his legal representative authorized by the patient signs the informed consent, fully understands the test content, process and possible adverse reactions, and is willing to follow up within the time specified in the test;
  2. Age 50-85 years old (including boundary value), male or female;
  3. The patient diagnosed with active choroidal neovascularization (CNV) disease secondary to wet age-related macular degeneration is confirmed by the reading center during screening;
  4. The total area of research eye lesions ≤ 30mm2 (12 optic disc areas), confirmed by the reading center before random enrollment;
  5. At the time of screening and baseline, the BCVA of the study eye was 73-24 letters (using the ETDRS visual acuity table, including the boundary value) (equivalent to the snellen visual acuity score of the study eye of 20/40 to 20/400);
  6. At the time of screening and baseline, the contralateral eye BCVA ≥ 34 letters (using the ETDRS visual acuity table, which is equivalent to snellen vision ≥ 20/200). For the subjects in the PK group, the investigator must judge that the contralateral eye is expected to be 3 No anti-VEGF treatment is required within a month.

Exclusion Criteria:

* If a patient meets any of the following conditions, they cannot enter the study:

Those with the following eye conditions:

1. The research eye has map-like atrophy involving the fovea, scars or fibrosis, anterior macular membrane, dense exudate hard exudation, RPE tear, etc. (confirmed by the reading center during screening);
2. Research eye retinal hemorrhage ≥ 4 optic disc areas (confirmed by the reading center during screening);
3. The research eye has significant interference with vision detection, anterior segment and fundus assessment of the refractive medium is turbid or the pupil is not dilated;
4. The research eye is combined with other fundus diseases (such as diabetic retinal degeneration, retinal vein occlusion, vascular streaking, pathological myopia, retinal detachment, macular hole, toxoplasmosis, optic nerve disease, etc.);
5. The research eye has pupil afferent defects (APD)
6. There are uncontrolled glaucoma in the research eye at the time of screening and baseline, defined as the intraocular pressure is still higher than 21mmHg after drug treatment, or according to the investigator's judgment;
7. The pre-screening research eye had received dexamethasone intravitreal implant (Ozurdex) treatment or fluocinolone intravitreal implant (Iluvien) treatment;
8. Within 3 months before the screening, the research eye had received the following treatments: photodynamic therapy (PDT), total retina laser photocoagulation, macular laser photocoagulation, transpupillary thermotherapy, etc., for AMD therapy;
9. The research eye has undergone the following ophthalmic operations: vitrectomy, macular transposition, anti-glaucoma surgery;
10. Have undergone external eye surgery or cataract surgery within 3 months before the study eye screening or during the study period;
11. The study eye has no lens (excluding intraocular lens) or posterior lens capsule rupture (except YAG laser posterior capsulotomy after implantation of intraocular lens more than 1 month after screening);
12. Contralateral eye received photodynamic (PDT) treatment within 1 month before screening;
13. A history of uveitis in any eye;
14. Vitreous hemorrhage in any eye during the screening period or history of vitreous hemorrhage within 4 weeks before baseline;
15. Any eye has pseudocapsular exfoliation syndrome;
16. Any eye has active eye infection (eg: blepharitis, infectious conjunctivitis, keratitis, scleritis, iridocyclitis, endophthalmitis);
17. Within 3 months before the screening, any eye had received intravitreal injection of anti-VEGF drugs (such as abecept, compaq, ranibizumab, bevacizumab, etc.);
18. Injection of corticosteroid drugs (such as triamcinolone acetonide, dexamethasone, etc.) into any eye, periocular or subconjunctival eye within 3 months before screening;

    Those with any of the following general conditions:
19. Currently in use or may need to use systemic drugs that may cause crystal toxicity or retinal toxicity, such as deferoxamine, chloroquine/hydroxychloroquine, phenothiazine, ethambutol or tamoxifen, etc.;
20. Have an allergic reaction or history of fluorescein sodium and indocyanine green, have a history of allergy to protein products for treatment or diagnosis, or are known to have allergic reactions to any monoclonal antibody;
21. Previously received systemic anti-VEGF treatment;
22. Patients with large doses of oral or injectable corticosteroids and other hormonal drugs (>10 mg prednisolone or the same dose/day) within 6 months before screening, but patients who use steroid drugs for inhalation, nasal cavity or local skin small doses except;
23. Poorly controlled diabetic patients are defined as glycated hemoglobin> 10%;
24. Those who had surgery within 1 month before screening and did not heal, or according to the judgment of the investigator;
25. There are clinically significant systemic infectious diseases that require intravenous antibiotic therapy;
26. Those who have a history of myocardial infarction, cerebral infarction and angina within 6 months before screening;
27. Those who have active disseminated intravascular coagulation and obvious bleeding tendency within 3 months before screening, or have received anticoagulant and antiplatelet therapy except aspirin/NSAIDs within 14 days before screening;
28. Hypertension patients with poor control (defined as blood pressure >160/100 mmHg after treatment with antihypertensive drugs);
29. Any uncontrollable clinical problems (such as severe mental, neurological, cardiovascular, respiratory and other system diseases and malignant tumors);

    Those with abnormalities in any of the following laboratory tests:
30. Abnormal liver and kidney function (this test stipulates that ALT and AST shall not be higher than the upper limit of the normal value of the laboratory in the center by 2.5 times; Crea and BUN shall not be higher than the upper limit of the normal value of the laboratory in the center by 2 times);
31. Patients with abnormal blood coagulation function (prothrombin time> upper limit of normal value 3 seconds or activated partial thromboplastin time> upper limit of normal value 10 seconds);
32. Any one of the following infected patients: active hepatitis B (if HBsAg(+) requires HBV DNA must be >500 IU/mL or the hospital maximum limit), hepatitis C, AIDS or syphilis (syphilis RPR positive test) ;

    Women and men of childbearing age in any of the following situations:
33. Women who are pregnant, pregnant or breastfeeding (pregnancy is defined as a positive blood/urine pregnancy test in this trial); male or female subjects of fertility do not agree to the entire study period and within 3 months after the end of the visit period Take appropriate contraceptive measures (such as IUDs, birth control pills or condoms, etc.). For women who have not been menopausal or have been menopausal but have not met the menopause time continuously for more than 12 months, and have not undergone sterilization surgery (ovarian and/or hysterectomy), they are defined as having fertility. The definition of fertility may be adjusted according to local standards in each region.

    Note: High-efficiency contraception methods include total abstinence, IUD, double barrier method (eg condom + diaphragm with spermicides, implanted contraceptives, hormonal contraceptives [contraceptives, implanted contraceptives, transdermal Patches, hormone-vaginal appliances or sustained-release injections], or the partner has undergone vasectomy and is confirmed to have no sperm); other:
34. Those who have participated in clinical trials of any drugs (excluding vitamins and minerals) within 3 months before screening;
35. The researchers believe that those who need to be excluded.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Dose-response relationships | week 24
  Trend chart of changes in the best corrected visual acuity from baseline

SECONDARY OUTCOMES:
BCVA | week 12 ，week 48
  the best corrected visual acuity
CRT | week 12 ，week 24，week 48
  The mean thickness of the central retina with a diameter of 1mm, centered on the fixed point of view
95% confidence interval | week 12 ，week 24，week 48
  The estimated interval of the population parameters constructed from the sample statistics
Average times of administration | week 24，week 48
  The times of administration of each dose group were summarized

OTHER OUTCOMES:
Pharmacokinetic（Cmax） | up tp week 48
  Pharmacokinetic parameters
Pharmacokinetic（Tmax） | up tp week 48
  Pharmacokinetic parameters
Pharmacokinetic（AUC0-Tau） | up tp week 48
  Pharmacokinetic parameters
Pharmacokinetic（AR） | up tp week 48
  Pharmacokinetic parameters
Pharmacokinetic（DF） | up tp week 48
  Pharmacokinetic parameters
Pharmacokinetic（t1/2） | up tp week 48
  Pharmacokinetic parameters
Pharmacokinetic（Vz） | up tp week 48
  Pharmacokinetic parameters
Pharmacokinetic（Vss） | up tp week 48
  Pharmacokinetic parameters
Pharmacokinetic（CL） | up tp week 48
  Pharmacokinetic parameters
VEGF | up tp week 48
  Peripheral vascular endothelial growth factor analysis
ADA | up tp week 48
  Immunogenicity analysis

CONTACTS AND LOCATIONS:
Overall Officials: Youxin Chen, Principal Investigator — Peking Union Medical College
Locations (16):
- China (16):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Eye Hospital of China Academy of Chinese Medical Sciences, Beijing
  - Peking University First Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Jieyang People's Hospital, Jieyang
  - The First Hospital of Jilin University, Jilin
  - he Affiliated Eye Hospital of Nanchang University, Nanchang
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Joint Shantou International Eye Center of Shantou University and The Chinese University of Hong Kong, Shantou
  - West China Hospital of Sichuan University, Sichuan
  - Wenzhou Medical University Affiliated Optometry Hospital, Wenzhou
  - The Second Xiangya Hospital of Central South University, Xiangya
  - Henan Provincial Eye Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided